CLINICAL TRIAL: NCT05693272
Title: A Randomized, Observer-Blind, Dose Escalation, Placebo-Controlled, Phase 1 Clinical Trial to Study the Safety and Immunogenicity of a COVAC-1 Booster Dose in Generally Healthy Adults
Brief Title: A Clinical Trial to Study the COVAC-1 Booster Dose in Generally Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Government of Canada (Other Government); Government of Saskatchewan (Other Government)
Responsible Party: Principal Investigator, Volker Gerdts, Director & CEO Vaccine and Infectious Disease Organization, University of Saskatchewan
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVAC-005
Record Dates: First submitted 2022-12-22; First posted 2023-01-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 Infection
Keywords: COVID-19 Booster Vaccine
MeSH Terms: conditions — COVID-19 | interventions — COVAC-1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COVAC-01 10µg group (Experimental): 12 healthy adults ≥18 years of age receive the vaccine on Day 0.
  Interventions: Biological: COVAC-1
- COVAC-01 25µg group (Experimental): 12 healthy adults ≥18 years of age receive the vaccine on Day 0.
  Interventions: Biological: COVAC-1
- COVAC-01 50µg group (Experimental): 12 healthy adults ≥18 years of age receive the vaccine on Day 0.
  Interventions: Biological: COVAC-1
- Placebo Control (Placebo Comparator): 12 healthy adults ≥18 years of age receive a dose of normal saline (placebo) on Day 0.
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: COVAC-1 — Intramuscular vaccine against SARS-CoV-2
  Arms: COVAC-01 10µg group; COVAC-01 25µg group; COVAC-01 50µg group
Biological: Saline Placebo — Intramuscular injection of saline placebo
  Arms: Placebo Control

SUMMARY:
VIDO has developed a vaccine called COVAC-1.

The COVAC-1 study vaccine contains a portion of the SARS-CoV-2 spike protein, called S1. The spike protein is the part of the virus that is responsible for attaching to the surface of host cells. COVAC-1 contains a TriAdj adjuvant. An adjuvant is a compound that is added to a vaccine to help the vaccine produce a better immune response. The vaccine is expected to stimulate the body to make antibodies against the S1 protein. The antibodies will recognize the viral spike protein if the body is exposed to the virus and prevent COVID-19 illness. In animal studies, the immune response generated by the COVAC-1 vaccine was able to protect the vaccinated animals against a severe SARS-CoV-2 infection.

The COVAC-005 Study is a Phase I, multi-centre trial of a SARS-CoV-2 vaccine booster. This is a randomized, observer-blinded, and placebo-controlled study to assess the safety and immunogenicity of COVAC-1 booster dose administered once in generally healthy adults 18-65 years of age who have received a minimum of 2 doses of an authorized COVID-19 vaccine at least 4 months prior to Day 0.

The study will follow a dose-escalation design to test the safety and immunogenicity of three dosage levels (10, 25 and 50 µg). In each dose escalation group participants will be randomized in a 3:1 ratio, to receive either the investigational product or a placebo, respectively. Stratification will be according to the Investigational product dose received. Sub-analysis will be completed in two age groups, 18-54 and 55-65 years.

Study participants will be initially randomized to the lowest dose of 10 µg or placebo. After approval by the Sponsor and based on the recommendations from the DSMB following the Day 7 safety analysis, new study participants will be allowed to be randomized in the higher dose escalation group of 25 µg. Approval will also be sought from the Sponsor, based upon the DSMB recommendation, to proceed with the higher dose of 50 µg. Within each dose escalation group of 16 participants (12 active vaccine recipients, and 4 placebo recipients) it is proposed to randomize a first cohort of 4 participants, including at least 3 active vaccine recipients, and pending no holding rule is met after 48 hours, as determined by the post-injection phone call, the remaining 12 participants within that dose escalation group will be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18-65 years of age at the time of signing the informed consent form for the study.
2. Good general health as confirmed by assessments completed no more than 30 days before study D0. Participants with mild to moderate well controlled comorbidities or having a medically stable condition, will be eligible. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization due to worsening during the 3 months prior to enrollment, and according to the judgment of the Investigator, hospitalization during the entire study period is not anticipated.
3. Have received a minimum of 2 doses of an authorized COVID-19 vaccine at least 4 months prior to the investigational booster dose injection. Proof of vaccination can be provided as a digital copy of the vaccination receipt on the participant's device, a screenshot of the receipt on the device, or a printed paper copy.
4. Male participants, and heterosexually active females of child-bearing potential, must practice adequate contraception for 30 days prior to the injection and must agree to continue adequate contraception until 180 days after the injection. Negative pregnancy test will be obtained from female participants of child-bearing potential at screening and at Day 0.
5. Provide a written informed consent for the study prior to performing any study-related procedure. The Investigator or a qualified designee must ensure the appropriate consent is in place.

Exclusion Criteria:

1. Presence of any febrile illness or any known or suspected acute illness on the day of immunization.
2. Clinically significant bleeding disorder (e.g., clotting factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injection or venipuncture.
3. Presence of an autoimmune disease.
4. Receiving systemic steroids in doses exceeding 20mg daily of prednisone or equivalent, for ≥ 14 days within 1 month, or has recently received any other cytotoxic or immunosuppressive drug within 6 months prior to the injection of the study vaccine.
5. Has a known malignancy diagnosed within the past 5 years. Participants with basal cell carcinoma or squamous cell carcinoma of the skin are not excluded.
6. Currently receiving systemic immunomodulatory therapy or received chemotherapy within the last 5 years excluding topical agents.
7. Has received blood products or immunoglobulins (IVIg or IMIg) within 3 months of study entry/baseline serologic evaluation.
8. Currently on anti-tuberculosis therapy.
9. Had SARS-CoV-2 infection within 4 months prior to study Day 0. A potential participant is considered to have COVID-19 infection base on one of the following:

   * Positive polymerase chain reaction (PCR) or rapid antigen test.
   * Documentation in a medical history report.
   * Reported by candidate.
10. Has received any non-COVID-19 authorized vaccines (e.g., influenza) within 2 weeks prior to receiving study dose injection.
11. Has received any experimental SARS-CoV-2 / COVID-19 vaccines Receipt of SARSCoV-2/COVID-19 vaccines that were experimental at the time of administration but are currently authorized, more than 6 months prior to Day 0, will not lead to exclusion.
12. Planning to receive booster doses of any authorized COVID-19 vaccine during the first two months days from study vaccination.
13. Abnormal laboratory test results (hematology, biochemistry, and urinalysis) as compared to the local normal lab ranges. To exclude transient abnormalities, laboratory tests may be repeated once. Abnormal lab test results considered not clinically significant by the Investigator will not be exclusionary.
14. Has a history of any reaction or known sensitivity likely to be exacerbated by any component of the study vaccine.
15. Is currently participating in or has participated in a study of an investigational agent within 6 months prior to the injection of the booster vaccine under study.
16. A female is not eligible to participate if she is pregnant or breast feeding
17. Being a member of the study team, or an immediate family member or household member of a member on the study team.
18. Any condition, which in the opinion of the investigator may deem the participant inappropriate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety of COVAC-1 booster vaccine (10, 25 and 50 μg dosing of S1 antigen) in generally healthy volunteers | Up to 365 days
  Incidence of solicited adverse events (AE) up to 7 days post-injection; unsolicited AEs up to 28 days post-injection; any clinically significant laboratory finding up to 28 days post-injection; and any serious AEs (SAEs), potential immune medicated disease (pIMDs), medically attended events or COVID-19 illness up to 365 days.

SECONDARY OUTCOMES:
To assess the antibody response induced by COVAC-1 booster pre-injection and post injection as measured by spike protein-specific Enzyme Linked Immunosorbent Assay (ELISA) | Up to Day 365.
  Study samples will be tested to assess the level of anti-SARS-CoV-2 spike IgG binding antibodies present in the human serum samples by using a validated ELISA.
To assess the immune response induced by COVAC-1 booster vaccine, as measured by cell immune response markers using flow cytometry. | Up to Day 365.
  Peripheral Blood Mononuclear Cells (PBMCs) samples collected pre- and post-injection will be assessed for spike protein-specific Helper T-lymphocytes (CD4+) and Cytotoxic T-lymphocytes (CD8+) population producing cytokine profile.
To assess the immune response induced by COVAC-1 booster vaccine, as measured by cell immune response markers using an ELISpot assay. | Up to Day 365.
  Peripheral Blood Mononuclear Cells (PBMCs) samples collected pre- and post-injection will be assessed for spike peptide-specific T cell responses, IFN-gamma and IL-5, as a measurement of COVAC-1 immune response induction.
To assess the antibody response induced by COVAC-1 booster pre-injection and post injection as measured by virus microneutralization assay. | Up to Day 365.
  Study samples will be tested to assess the level of SARS-CoV-2 Wuhan neutralizing antibodies present in the human serum samples by SARS-CoV-2 live virus microneutralization assay.
To assess the antibody response induced by COVAC-1 booster pre-injection and post injection as measured by pseudovirus neutralization assay. | Up to Day 365.
  Study samples will be tested to assess the level of SARS-CoV-2 Wuhan pseudovirus neutralizing antibodies present in the human serum samples by SARS-CoV-2 pseudotyped virus neutralization assay.

OTHER OUTCOMES:
To assess the neutralizing antibody response induced by COVAC-1 against the Omicron and/or the most relevant currently circulating Variants of Concern. | Up to 365 days
  Study samples will be tested to assess the level of neutralizing antibodies against the SARS-CoV-2 Omicron Variant of Concern and/or against other currently circulating Variants of Concern, present in the human serum samples by SARS-CoV-2 live virus microneutralization assay.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Diex Recherche Joliette Inc., Joliette, Quebec
  - Diex Recherche Quebec Inc., Québec, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - DIEX Recherche Victoriaville, Victoriaville, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garg R, Liu Q, Van Kessel J, Asavajaru A, Uhlemann EM, Joessel M, Hamonic G, Khatooni Z, Kroeker A, Lew J, Scruten E, Pennington P, Deck W, Prysliak T, Nickol M, Apel F, Courant T, Kelvin AA, Van Kessel A, Collin N, Gerdts V, Koster W, Falzarano D, Racine T, Banerjee A. Efficacy of a stable broadly protective subunit vaccine platform against SARS-CoV-2 variants of concern. Vaccine. 2024 Aug 13;42(20):125980. doi: 10.1016/j.vaccine.2024.05.028. Epub 2024 May 19. PMID 38769033